CLINICAL TRIAL: NCT01034137
Title: U-ACT-EARLY: A Multi-center, Randomized, Double Blind, Placebo Controlled Study to Evaluate Remission in DMARD and Biological naïve Early Rheumatoid Arthritis (RA) Subjects Treated With Tocilizumab (TCZ) Plus Tight Control Methotrexate (MTX) , TCZ Monotherapy or Tight Control MTX Monotherapy
Brief Title: A Study of Tocilizumab and Methotrexate in Combination or as Monotherapy in Treatment-Naïve Patients With Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML22497; 2009-013316-12
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Treat-to-target, tight control, strategy study, TCZ, MTX
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tocilizumab + Methotrexate (Experimental): Participants will receive intravenous (IV) TCZ 8 mg/kg every four weeks for a maximum of 26 infusions + oral capsules of MTX 10-30 mg/week in climbing dosages of 5 mg starting at 10 mg up till a maximum dosage of 30 mg/week. The weekly dose of MTX will be taken on one particular day of the week.
  Interventions: Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]
- Tocilizumab + Placebo Methotrexate (Active Comparator): Participants will receive IV TCZ 8 mg/kg every four weeks for a maximum of 26 infusions + weekly oral matching placebo MTX capsules in climbing dosages. The weekly dose of placebo MTX will be taken on one particular day of the week.
  Interventions: Drug: placebo MTX; Drug: tocilizumab [RoActemra/Actemra]
- Methotrexate + Placebo Tocilizumab (Active Comparator): Participants will receive weekly oral MTX in climbing dosages of 5 mg starting at 10 mg up till a maximum dosage of 30 mg/week + matching placebo TCZ IV 8 mg/kg every four week for a maximum of 26 infusions. The weekly dose of MTX will be taken on one particular day of the week.
  Interventions: Drug: methotrexate; Drug: placebo TCZ

INTERVENTIONS:
Drug: methotrexate — orally weekly in ascending dosages, starting at 10mg/week
  Arms: Methotrexate + Placebo Tocilizumab; Tocilizumab + Methotrexate
Drug: placebo MTX — orally weekly
  Arms: Tocilizumab + Placebo Methotrexate
Drug: placebo TCZ — iv every 4 weeks
  Arms: Methotrexate + Placebo Tocilizumab
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks
  Arms: Tocilizumab + Methotrexate; Tocilizumab + Placebo Methotrexate

SUMMARY:
This randomized, double-blind, placebo-controlled study will compare the efficacy with regard to sustained remission and safety of tocilizumab and methotrexate, in combination or as monotherapy, in treatment-naïve patients with early rheumatoid arthritis. Patients will be randomized to receive either tocilizumab (8mg/kg iv every 4 weeks) plus weekly methotrexate (po in ascending doses), or tocilizumab (8mg/kg iv every 4 weeks) plus placebo, or methotrexate plus placebo. Anticipated time on study treatment is 2 years, and target sample size is 300.

DETAILED DESCRIPTION:
Multi-center, randomized, double-blind, placebo-controlled (double placebo) three-arm parallel group, comparative study. Patients were randomized in a 1:1:1 ratio to one of the following treatments:

* TCZ 8 milligram (mg)/kilogram (kg) + MTX (Group I: TCZ+MTX)
* TCZ 8 mg/kg + placeboMTX (Group II: TCZ+placebo)
* MTX + placeboTCZ (Group III: MTX+placebo)

Randomization was stratified by participating center and baseline Disease Activity Score, scoring 28 joints (DAS28) level (<5.1 vs. ≥5.1). Patients were evaluated every 4 weeks and at each visit a decision on dosage changes was made based on efficacy parameters (DAS28) and occurrence of adverse events (AEs). Patients received MTX/placeboMTX in climbing dosages. Hydroxychloroquine (HCQ) was added when remission was not reached with the maximum tolerable dosage (MTD) of MTX/placeboMTX. If after 12 additional weeks remission was not reached, HCQ was stopped and replaced by standard of care therapy (in Group I) or placebo therapy was replaced by the corresponding verum resulting in TCZ+MTX combination therapy (in Groups II and III). In case remission was reached, MTX/placeboMTX and TCZ/placeboTCZ had to be decreased. Patients were followed for a maximum of 24 months

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* early rheumatoid arthritis (disease symptoms <1 year) according to ACR criteria
* disease activity DAS28 >2.6
* body weight </=110kg, BMI </=36

Exclusion Criteria:

* rheumatic autoimmune disease other than RA
* current inflammatory joint disease other than RA
* previous treatment with any DMARD or biologic drug used in the treatment of RA
* intra-articular, parenteral or oral glucocorticoids used for the arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2010-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Netherlands (21):
  - Alkmaar
  - Amersfoort
  - Amsterdam
  - Apeldoorn
  - Breda
  - Den Helder
  - Emmeloord
  - Gorinchem
  - Gouda
  - Groningen
  - Haarlem
  - Heerlen
  - Hilversum
  - Hoofddorp
  - Leeuwarden
  - Leiden
  - Nieuwegein
  - Nijmegen
  - Sneek
  - Utrecht
  - Woerden

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gosselt HR, Verhoeven MMA, de Rotte MCFJ, Pluijm SMF, Muller IB, Jansen G, Tekstra J, Bulatovic-Calasan M, Heil SG, Lafeber FPJG, Hazes JMW, de Jonge R. Validation of a Prognostic Multivariable Prediction Model for Insufficient Clinical Response to Methotrexate in Early Rheumatoid Arthritis and Its Clinical Application in Evidencio. Rheumatol Ther. 2020 Dec;7(4):837-850. doi: 10.1007/s40744-020-00230-7. Epub 2020 Sep 14. PMID 32926395
- [Derived] Teitsma XM, Yang W, Jacobs JWG, Petho-Schramm A, Borm MEA, Harms AC, Hankemeier T, van Laar JM, Bijlsma JWJ, Lafeber FPJG. Baseline metabolic profiles of early rheumatoid arthritis patients achieving sustained drug-free remission after initiating treat-to-target tocilizumab, methotrexate, or the combination: insights from systems biology. Arthritis Res Ther. 2018 Oct 15;20(1):230. doi: 10.1186/s13075-018-1729-2. PMID 30322408
- [Derived] Teitsma XM, Jacobs JWG, Welsing PMJ, de Jong PHP, Hazes JMW, Weel AEAM, Petho-Schramm A, Borm MEA, van Laar JM, Lafeber FPJG, Bijlsma JWJ. Inadequate response to treat-to-target methotrexate therapy in patients with new-onset rheumatoid arthritis: development and validation of clinical predictors. Ann Rheum Dis. 2018 Sep;77(9):1261-1267. doi: 10.1136/annrheumdis-2018-213035. Epub 2018 May 14. PMID 29760159
- [Derived] Teitsma XM, Jacobs JWG, Welsing PMJ, Petho-Schramm A, Borm MEA, van Laar JM, Lafeber FPJG, Bijlsma JWJ. Radiographic joint damage in early rheumatoid arthritis patients: comparing tocilizumab- and methotrexate-based treat-to-target strategies. Rheumatology (Oxford). 2018 Feb 1;57(2):309-317. doi: 10.1093/rheumatology/kex386. PMID 29095992
- [Derived] Teitsma XM, Jacobs JWG, Welsing PMJ, Petho-Schramm A, Borm MEA, Hendriks L, Denissen NHAM, van Laar JM, Lafeber FPJG, Bijlsma JWJ. Patient-reported outcomes in newly diagnosed early rheumatoid arthritis patients treated to target with a tocilizumab- or methotrexate-based strategy. Rheumatology (Oxford). 2017 Dec 1;56(12):2179-2189. doi: 10.1093/rheumatology/kex319. PMID 29029185
- [Derived] Teitsma XM, Jacobs JWG, Mokry M, Borm MEA, Petho-Schramm A, van Laar JM, Bijlsma JWJ, Lafeber FPJ. Identification of differential co-expressed gene networks in early rheumatoid arthritis achieving sustained drug-free remission after treatment with a tocilizumab-based or methotrexate-based strategy. Arthritis Res Ther. 2017 Jul 20;19(1):170. doi: 10.1186/s13075-017-1378-x. PMID 28728565
- [Derived] Bijlsma JWJ, Welsing PMJ, Woodworth TG, Middelink LM, Petho-Schramm A, Bernasconi C, Borm MEA, Wortel CH, Ter Borg EJ, Jahangier ZN, van der Laan WH, Bruyn GAW, Baudoin P, Wijngaarden S, Vos PAJM, Bos R, Starmans MJF, Griep EN, Griep-Wentink JRM, Allaart CF, Heurkens AHM, Teitsma XM, Tekstra J, Marijnissen ACA, Lafeber FPJ, Jacobs JWG. Early rheumatoid arthritis treated with tocilizumab, methotrexate, or their combination (U-Act-Early): a multicentre, randomised, double-blind, double-dummy, strategy trial. Lancet. 2016 Jul 23;388(10042):343-355. doi: 10.1016/S0140-6736(16)30363-4. Epub 2016 Jun 7. PMID 27287832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 360 participants were screened at 21 centers in the Netherlands from 04 JAN 2010 to 30 JUL 2012.
Pre-assignment Details: Of 360 participants, 43 failed screening.
Groups:
- Tocilizumab + Methotrexate: Participants received intravenous (IV) Tocilizumab (TCZ) 8 milligram (mg)/kilogram (kg) every four weeks for a maximum of 26 infusions + oral capsules of Methotrexate (MTX) 10-30 mg/week in climbing dosages of 5 mg starting at 10 mg up till a maximum dosage of 30 mg/week. The weekly dose of MTX was taken on one particular day of the week.
- Tocilizumab + Placebo Methotrexate: Participants received IV TCZ 8 mg/kg every four weeks for a maximum of 26 infusions + weekly oral matching placebo MTX capsules in climbing dosages. The weekly dose of placebo MTX was taken on one particular day of the week.
- Methotrexate + Placebo Tocilizumab: Participants received weekly oral MTX in climbing dosages of 5 mg starting at 10 mg up till a maximum dosage of 30 mg/week + matching placebo TCZ IV 8 mg/kg every four week for a maximum of 26 infusions. The weekly dose of MTX was taken on one particular day of the week.
Period: Overall Study
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Started | 106 | 103 | 108
Completed | 78 | 81 | 78
Not Completed | 28 | 22 | 30
Not completed — Adverse Event | 9 | 10 | 8
Not completed — Withdrawal by Subject | 4 | 3 | 3
Not completed — Lack of Efficacy | 9 | 4 | 13
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Refused treatment or did not cooperate | 2 | 0 | 1
Not completed — Administrative or other | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab + Methotrexate: Participants received IV TCZ 8 mg/ kg every four weeks for a maximum of 26 infusions + oral capsules of MTX 10-30 mg/week in climbing dosages of 5 mg starting at 10 mg up till a maximum dosage of 30 mg/week. The weekly dose of MTX was taken on one particular day of the week.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab | Total
Number analyzed (Participants) | 106 | 103 | 108 | 317
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 85 | 79 | 87 | 251
  >=65 years | 21 | 24 | 21 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (11.8) | 55.0 (12.9) | 52.2 (13.7) | 53.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 78 | 69 | 212
  Male | 41 | 25 | 39 | 105

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Remission Rate At Week 104
Description: Sustained remission rate (SRR) is defined as Disease Activity Score 28 (DAS28) <2.6 during ≥ 23 weeks and no more than 4 swollen joints (28 joint count) due to RA at Week 24 of remission, with the exception of up to 2 in-between DAS28 values which could be between 2.6 and 3.2. The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores indicate worsening. DAS28 <2.6 equals (=) remission.
Time Frame: Week 104
Population: The intent to treat (ITT) population consisted of all participants who were randomized and received at least one dose of TCZ/placebo infusion or MTX/placebo capsules and performed at least one post-baseline efficacy measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Percentage of participants | 85.8 | 83.5 | 44.4
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Methotrexate + Placebo Tocilizumab; The SRR was compared between the treatment groups by means of the Cochran-Mantel-Haenszel (CMH) test taking into account the stratification factors used for randomization; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.996, 95% CI 2-sided [1.589 to 2.506]
Statistical Analysis 2: Comparison: Tocilizumab + Placebo Methotrexate vs Methotrexate + Placebo Tocilizumab; The SRR was compared between the treatment groups by means of the CMH test taking into account the stratification factors used for randomization; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.855, 95% CI 2-sided [1.481 to 2.323]
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo Methotrexate; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.616, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.030, 95% CI 2-sided [0.915 to 1.160]

2. Secondary Outcome: Median Time to First Sustained Remission
Description: It is the time to event analysis for the first period of sustained remission. Sustained remission is defined as DAS28 <2.6 during ≥23 weeks and no more than 4 swollen joints (28 joint count) due to RA at Week 24 of remission, with the exception of up to 2 in-between DAS28 values which could be between 2.6 and 3.2. The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen and tender joint counts (range 0-28), acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores indicate worsening. DAS28 <2.6 equals (=) remission.
Time Frame: Up to Week 104
Population: The ITT population consisted of all participants who were randomized and received at least one dose of TCZ/placebo infusion or MTX/placebo capsule and performed at least one post-baseline efficacy measurement.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
days | 69.00 [57.00 to 85.00] | 89.00 [58.00 to 116.00] | NA [243.00 to NA] — As there was not that much sustained remission in the MTX + PBO group, median time to remission could not be calculated.

3. Secondary Outcome: Mean Duration of First Sustained Remission
Description: It is the duration of the first period of sustained DAS28 remission. Participants who switch treatment strategy before reaching sustained remission considered failures.
Time Frame: Up to Week 104
Population: The ITT population consisted of all participants who were randomized and received at least one dose of TCZ/placebo infusion or MTX/placebo capsule and performed at least one post-baseline efficacy measurement. n = number of participants evaluable at particular time of assessment.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 91 | 86 | 48
Weeks | 65.85 (26.70) | 65.00 (24.75) | 52.90 (25.11)

4. Secondary Outcome: Number of Participants Achieving Disease Activity Score 28 Remission at Weeks 12, 24, 52, and 104
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores indicate worsening. DAS28 <2.6 equals (=) remission. Participants with missing data at visits before early study termination or who stopped the study prematurely because of insufficient therapeutic response or safety reasons considered non-responders or who stopped the study for other reasons, response set to missing after early withdrawal.
Time Frame: Weeks 12, 24, 52, and 104
Population: as for outcome 3
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 105 | 102 | 106
Number of participants
  Week 12, n=105, 102, 106 | 76 | 66 | 23
  Week 24, n=105, 102, 106 | 84 | 77 | 42
  Week 52, n=100, 99, 103 | 71 | 80 | 63
  Week 104, n=96, 95, 99 | 71 | 67 | 58

5. Secondary Outcome: Median Time to First Disease Activity Score 28 Remission
Description: It is the time to event analysis for the first DAS28 remission.
Time Frame: Up to Week 104
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Days | 56.00 [54.00 to 58.00] | 57.00 [49.00 to 60.00] | 167.00 [138.00 to 195.00]

6. Secondary Outcome: Percentage of Participants With Cumulative Remission Rate at Weeks 12, 24, 52, and 104
Description: The DAS28 score is a measure of the subject's disease activity. DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement. Participants with missing data at visits before early study termination or who stopped the study prematurely because of insufficient therapeutic response or safety reasons considered non-responders or who stopped the study for other reasons, response set to missing after early withdrawal.
Time Frame: Weeks 12, 24, 52, and 104
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 105 | 102 | 106
Percentage of participants
  Week 12, n=105,102,106 | 72.4 | 64.7 | 21.7
  Week 24, n=105,102,106 | 80.0 | 75.5 | 39.6
  Week 52, n=100, 99,103 | 71.0 | 80.8 | 61.2
  Week 104, n=96, 95, 99 | 63.5 | 70.5 | 58.6

7. Secondary Outcome: Mean Duration of First Disease Activity Score 28 Remission
Description: It is the duration of the first period of DAS28 remission.
Time Frame: Up to Week 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Weeks | 42.99 (31.79) | 37.01 (30.89) | 20.49 (23.95)

8. Secondary Outcome: Absolute Change From Baseline in Disease Activity Score 28 at Weeks 12, 24, 52, and 104
Description: The DAS28 score is a measure of the participant's disease activity. DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement. Participants with missing data at visits before early study termination or who stopped the study prematurely because of insufficient therapeutic response or safety reasons considered non-responders or who stopped the study for other reasons, response set to missing after early withdrawal.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52, and 104
Population: as for outcome 2
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Scores on a scale
  Week 12 | 3.1 [-0.21 to 7.34] | 3.3 [0.37 to 6.76] | 1.4 [-1.53 to 3.91]
  Week 24 | 3.6 [0.75 to 7.48] | 3.6 [0.45 to 7.64] | 2.1 [-1.67 to 5.11]
  Week 52 | 3.3 [-1.02 to 7.48] | 3.4 [0.28 to 7.66] | 3.3 [-0.74 to 6.13]
  Week 104 | 3.3 [-0.73 to 6.07] | 3.3 [0.1 to 6.8] | 3.2 [-0.79 to 7.52]

9. Secondary Outcome: Median Change From Baseline in Clinical Disease Activity Index Score at Weeks 24, 52, and 104
Description: The clinical disease activity index (CDAI) are continuous measures of RA disease activity. The CDAI is the numerical sum of four outcome parameters: tender joint count (TJC), swollen joint count (SJC) based on a 28-joint assessment; and patient's global assessment (PtGA) and physician's global assessment (PhGA) assessed on 0-10 cm visual analog scale (VAS). CDAI total score ranges from 0 to 76. CDAI <= 2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high (or severe) disease activity.
Time Frame: From Baseline (Week 0) to Weeks 24, 52, and 104
Population: as for outcome 2
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Scores on a scale
  Week 24 | -20.0 [-66.5 to -1.5] | -20.0 [-62.5 to 13] | -14.8 [-42 to 13]
  Week 52 | -19.5 [-67 to 3] | -21.0 [-62.5 to 2] | -18.0 [-47.5 to -0.5]
  Week 104 | -19.0 [-39 to 6] | -21.5 [-62.5 to -1] | -18.0 [-51 to 12]

10. Secondary Outcome: Median Change From Baseline in Simplified Disease Activity Index Scores at Weeks 24, 52, and 104
Description: The simplified disease activity index (SDAI ) are continuous measures of RA disease activity.The SDAI is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PhGA (assessed on 0-10 cm VAS), and C-Reactive Protein (CRP) (mg/dL). SDAI total score ranges from 0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: From Baseline (Week 0) to Weeks 24, 52, and 104
Population: as for outcome 2
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Scores on a scale
  Week 24 | -31.0 [-282 to 6.4] | -32.8 [-290 to 12.1] | -21.5 [-186 to 45.5]
  Week 52 | -26.3 [-272.5 to 30] | -33.5 [-288 to 1.2] | -27.9 [-189 to -1.5]
  Week 104 | -25.6 [-98.9 to 11] | -32.8 [-293.5 to 6.5] | -28.0 [-188.4 to 14.9]

11. Secondary Outcome: Number of Participants With Good European League Against Rheumatism Response Rate at Weeks 24, 52, and 104
Description: European league against rheumatism (EULAR) response criteria classify each participant as a good, moderate or non-responder to treatment based on the degree of improvement from baseline and the level of disease activity at the endpoint. EULAR response is derived using the individual participant's DAS28 as the measure of severity of disease. Good or moderate response is defined as follows: Good response : DAS28 at the time point =<3.2 and improvement from baseline > 1.2. Moderate response : DAS28 at the time point > 3.2 and improvement from baseline > 1.2, or DAS28 at the time point ≤ 5.1 and improvement from baseline > 0.6 and =<1.2.
Time Frame: Weeks 24, 52, and 104
Population: as for outcome 3
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 105 | 97 | 103
Number of participants
  Week 24, n=105, 97, 103 | 93 | 84 | 50
  Week 52, n=100, 96, 99 | 75 | 85 | 71
  Week 104, n=96, 95, 96 | 63 | 72 | 65

12. Secondary Outcome: Median Time to First European League Against Rheumatism Response
Description: It is the time to first EULAR response. EULAR response criteria classify each participant as a good, moderate or non-responder to treatment based on the degree of improvement from baseline and the level of disease activity at the endpoint. EULAR response is derived using the individual participant's DAS28 as the measure of severity of disease.Good or moderate response is defined as follows: Good response : DAS28 at the time point ≤ 3.2 and improvement from baseline > 1.2. Moderate response : DAS28 at the time point > 3.2 and improvement from baseline > 1.2, or DAS28 at the time point ≤ 5.1 and improvement from baseline > 0.6 and ≤ 1.2. Response 1 is defined as yes (good) versus no (moderate or no response). Response 2 is defined as yes (good or moderate) versus no (no response).
Time Frame: Up to Week 104
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Days
  EULAR response 1 | 35.5 [29.0 to 58.0] | 47.0 [29.0 to 60.] | 132.0 [84.0 to 195.0]
  EULAR response 2 | 29.0 [28.0 to 30.0] | 29.0 [27.0 to 31.0] | 57.0 [29.0 to 85.0]

13. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20 Response Rate at Weeks 12, 24, 52 and 104
Description: American College of Rheumatology (ACR) 20 response is defined as a >= 20% improvement (reduction) compared with baseline for both tender joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: patient's assessment of pain over the previous 24 hours: using a Visual Analog Scale (VAS) with left end of the line 0=no pain to right end of the line 100=unbearable pain; patient's global assessment of disease activity and physician's global assessment of disease activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: Weeks 12, 24, 52 and 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Percentage of participants
  Weeks 12 | 63.8 | 67.6 | 41.5
  Weeks 24 | 75.2 | 75.5 | 59.4
  Weeks 52 | 74.7 | 71.7 | 68.9
  Weeks 104 | 63.5 | 65.3 | 60.6

14. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50 Response Rate at Weeks 12, 24, 52 and 104
Description: ACR50 response is defined as a >=50% improvement (reduction) compared with baseline for both TJC68 and SJC66, as well as for three of the additional five ACR core set variables: patient's assessment of pain over the previous 24 hours: using a VAS with left end of the line 0=no pain to right end of the line 100=unbearable pain; patient's Global assessment of disease activity and physician's global assessment of disease activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: Weeks 12, 24, 52 and 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Percentage of participants
  Week 12 | 47.6 | 44.1 | 21.7
  Week 24 | 63.8 | 58.8 | 34.0
  Week 52 | 61.6 | 58.6 | 51.5
  Week 104 | 49.0 | 54.7 | 48.5

15. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70 Response Rate at Weeks 12, 24, 52 and 104
Description: ACR70 response is defined as a >=70% improvement (reduction) compared with baseline for both TJC68 and SJC66, as well as for three of the additional five ACR core set variables: patient's Assessment of pain over the previous 24 hours: using a VAS with left end of the line 0=no pain to right end of the line 100=unbearable pain; patient's global assessment of disease activity and physician's global assessment of disease activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; health assessment questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: Weeks 12, 24, 52 and 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Percentage of participants
  Week 12 | 30.5 | 23.5 | 7.5
  Week 24 | 43.8 | 37.3 | 15.1
  Week 52 | 44.4 | 44.4 | 33.0
  Week 104 | 36.5 | 38.9 | 35.4

16. Secondary Outcome: Percentage of Participants With American College of Rheumatology 90 Response Rate at Weeks 12, 24, 52 and 104
Description: ACR90 response is defined as a >=90% improvement (reduction) compared with baseline for both tender joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a VAS with left end of the line 0=no pain to right end of the line 100=unbearable pain; patient's global assessment of disease activity and physician's global assessment of disease activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; health assessment questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or erythrocyte sedimentation rate.
Time Frame: Weeks 12, 24, 52 and 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Percentage of participants
  Weeks 12 | 9.5 | 3.9 | 0.0
  Weeks 24 | 18.1 | 11.8 | 4.7
  Weeks 52 | 19.2 | 21.2 | 6.8
  Weeks 104 | 20.8 | 20.0 | 14.1

17. Secondary Outcome: Mean Percent Change From Baseline in the Swollen Joint Count (SJC) at Weeks 12, 24, 52, and 104
Description: The number of swollen joints among 22 anatomical joints for both the right and left side of the body were assessed by a joint evaluator where the presence of a swollen joint was scored as 1 and absence as 0. The total SJC was derived by the sum of the scores for a range of SJC from 0 (best possible score; no swollen joints) to 44 (worse possible score; all joints swollen).
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52, and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 104 | 100 | 98
Percent change
  Week 12, n=104, 100, 98 | -69.2 (91.1) | -68.2 (45.1) | -44.9 (73.9)
  Week 24, n=100, 100, 97 | -91.7 (18.5) | -86.9 (24.3) | -69.3 (37.8)
  Week 52, n=86, 91, 87 | -93.3 (19.6) | -89.0 (24.1) | -91.3 (20.0)
  Week 104, n=78, 80, 77 | -85.7 (44.7) | -91.6 (31.3) | -87.9 (23.7)

18. Secondary Outcome: Mean Percent Change From Baseline in the Tender Joint Count (TJC) at Weeks 12, 24, 52, and 104
Description: The number of tender joints among 22 anatomical joints for both the right and left side of the body were assessed by a joint evaluator where the presence of a tender joint was scored as 1 and absence as 0. The total TJC was derived by the sum of the scores for a range of TJC from 0 (best possible score; no tender joints) to 44 (worse possible score; all tender joints).
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52, and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 102 | 98 | 99
Percent change
  Week 12, n=102, 98, 99 | -68.0 (44.6) | -53.7 (84.1) | -36.9 (65.9)
  Week 24, n=98, 98, 97 | -81.9 (28.8) | -66.1 (83.8) | -66.6 (34.0)
  Week 52, n=84, 89, 87 | -77.8 (49.8) | -80.4 (33.1) | -77.7 (33.6)
  Week 104, n=76, 79, 77 | -84.5 (26.4) | -82.5 (30.7) | -79.9 (31.9)

19. Secondary Outcome: Mean Percent Change From Baseline in Patient Health Visual Analog Scale at Weeks 12, 24, 52, and 104
Description: Patient health visual analog scale is a component of ACR. It is measured using a visual analogue scale with scores ranging from 0 to 100 (higher scores indicate worse disease activity). An improvement (decrease) in the patient's global assessment based on disease activity relative to respective baseline values was analyzed.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52, and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 96 | 97 | 97
Percent change
  Week 12, n =96, 97, 97 | -43.8 (75.2) | -40.8 (74.7) | -25.3 (69.0)
  Week 24, n=92, 96, 93 | -66.5 (36.5) | -54.8 (41.8) | -41.5 (62.4)
  Week 52, n=79, 82, 84 | -66.5 (37.7) | -63.4 (36.8) | -58.4 (69.6)
  Week 104, n=72, 72, 72 | -64.0 (39.7) | -67.4 (36.3) | -64.7 (39.2)

20. Secondary Outcome: Mean Percent Change From Baseline in The Physician Health Visual Analog Scale at Weeks 12, 24, 52, and 104
Description: Physician health visual analog scale is a component of ACR. It is measured using a visual analogue scale with scores ranging from 0 to 100 (higher scores indicate worse disease activity).An improvement (decrease) in the physician's global assessment based on disease activity parameter relative to respective baseline values was analyzed.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52, and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 104 | 101 | 100
Percent change
  Week 12, n =104, 101, 100 | -41.6 (47.2) | -36.5 (42.7) | -18.2 (52.5)
  Week 24, n =100, 101, 98 | -61.0 (37.7) | -46.7 (40.9) | -26.1 (57.9)
  Week 52, n =86, 92, 88 | -56.9 (42.8) | -56.2 (45.7) | -48.2 (50.1)
  Week 104, n =78, 81, 78 | -63.2 (37.0) | -60.2 (38.9) | -53.9 (54.8)

21. Secondary Outcome: Mean Percent Change From Baseline in Pain Visual Analog Scale at Weeks 12, 24, 52, and 104
Description: Pain VAS is a component of ACR. VAS pain score calculated as 0 to 10 cm; where 0 = no pain, and 10 = worst possible pain.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52, and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 82 | 83 | 77
Percent change
  Week 12, n=82, 83, 77 | -59.3 (37.6) | -55.8 (34.7) | -39.1 (43.5)
  Week 24, n=76, 77, 78 | -74.9 (31.4) | -70.3 (25.4) | -48.6 (52.6)
  Week 52, n=76, 72, 72 | -77.0 (30.9) | -72.4 (41.1) | -66.4 (35.9)
  Week 104, n=58, 61, 63 | -76.5 (35.0) | -78.8 (27.7) | -74.9 (27.3)

22. Secondary Outcome: Mean Percent Change From Baseline in CRP at Weeks 12, 24, 52, and 104
Description: CRP is a component of ACR. CRP is a marker of inflammation.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52, and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 103 | 101 | 100
Percent change
  Week 12, n=103, 101, 100 | -47.4 (216.5) | -69.8 (39.4) | -28.5 (65.9)
  Week 24, n=99, 101, 98 | -64.4 (72.1) | -69.1 (47.1) | -16.8 (127.7)
  Week 52, n=85, 92, 88 | -47.1 (107.2) | -51.9 (72.0) | -52.1 (100.4)
  Week 104, n=77, 81, 78 | -45.5 (105.8) | -12.7 (256.5) | -46.7 (65.5)

23. Secondary Outcome: Mean Change From Baseline in Modified Sharp/Van Der Heijde Score at Weeks 52 and 104
Description: The degree of joint damage was assessed using the van der Heijde modified total Sharp score (mTSS). The methodology quantifies the extent of bone erosions for 44 joints and joint space narrowing (JSN) for 42 joints, with higher scores representing greater damage. The independent read of X-ray images was performed by 2 primary readers. In case of discrepancy between the 2 primary readers, an adjudicator was involved. The mTSS can range from 0 to 448 with a higher score indicating more joint damage. A negative change score indicates improvement.
Time Frame: From Baseline (Week 0) to Weeks 52 and 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Scores on a scale
  Week 52 | 0.50 (1.495) | 0.79 (3.242) | 0.96 (2.870)
  Week 104 | 1.18 (3.919) | 1.45 (4.272) | 1.53 (2.421)

24. Secondary Outcome: Percentage of Participants Who Withdraw Due to Lack of Sufficient Therapeutic Response
Description: Insufficient therapeutic response (participants not responding to the drug as assessed by the physician) was selected by the investigator as a reason for the participant to withdraw from the study.
Time Frame: Up to Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Percentage of participants | 32.1 | 18.2 | 43.3

25. Secondary Outcome: Number of Participants With Change in The Therapy Strategy During The Study
Description: Participants who switched treatment strategy from monotherapy (TCZ+ placebo MTX or MTX+ placebo TCZ treatment) to combination therapy (TCZ+MTX treatment) was reported. Also, participants who switched from verum therapy to standard of care was reported in the below table.
Time Frame: From Baseline to Week 104
Population: as for outcome 2
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Number of participants
  Treatment strategy switch | 0 | 13 | 50
  Switch from verum to standard of care | 9 | 2 | 2

26. Secondary Outcome: Mean Change From Baseline in The Dutch Consensus Health Assessment Questionnaire of Quality of Life at Weeks 12, 24, 52, and 104
Description: The Dutch Consensus Health Assessment Questionnaire (DC-HAQ) disability index is a self-completed participant questionnaire with 8 domains specific for RA. It assesses a participant functional ability, with scores ranging from 0 (without any difficulty) to 3 (unable to do). A change from baseline of -0.22 is considered to be the minimal clinically important difference.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 95 | 95 | 91
Scores on a scale
  Week 12, n=95, 95, 91 | -0.5 (0.6) | -0.5 (0.5) | -0.2 (0.5)
  Week 24, n=92, 94, 87 | -0.7 (0.6) | -0.6 (0.6) | -0.4 (0.5)
  Week 52, n=81, 81, 82 | -0.7 (0.7) | -0.7 (0.6) | -0.5 (0.6)
  Weeks 104, n=68, 75, 71 | -0.6 (0.7) | -0.6 (0.6) | -0.4 (0.6)

27. Secondary Outcome: Mean Change From Baseline in The EuroQol Score of Quality of Life at Weeks 12, 24, 52 and 104
Description: "EuroQol (EQ-5D) is a standard self-completed participant questionnaire that measures health outcome. The EQ-5D questionnaire consists of 2 parts: 1) EQ-5D with five dimensions: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Each dimension is rated on a 3-point response scale as 1 = no problems, 2 = some/moderate problems, 3 = extreme problems. The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, where '1' indicating full health and '0' representing dead. The positive values indicate that during the study the health status improved. 2) EQ-VAS on a scale of 0 to 100, where 0 = worst possible health status and 100 = best possible health status."
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 72 | 73 | 78
Scores on a scale
  EQ-5D Week 12, n=72, 72, 78 | 0.15 (0.25) | 0.19 (0.25) | 0.11 (0.28)
  EQ-VAS Week 12, n=69, 70, 73 | 11.94 (21.07) | 9.31 (16.90) | 2.92 (17.54)
  EQ-5D Week 24, n=69, 73, 73 | 0.19 (0.22) | 0.15 (0.30) | 0.15 (0.27)
  EQ-VAS Week 24, n=67, 69, 71 | 13.15 (21.93) | 10.86 (21.46) | 8.97 (20.17)
  EQ-5D Week 52, n=61, 61, 69 | 0.18 (0.25) | 0.21 (0.24) | 0.25 (0.29)
  EQ-VAS Week 52, n=58, 59, 67 | 12.52 (21.61) | 13.71 (18.63) | 13.40 (24.45)
  EQ-5D Week 104, n=50,57,54 | 0.14 (0.22) | 0.20 (0.28) | 0.21 (0.29)
  EQ-VAS Week 104, n=50,52,57 | 10.88 (20.43) | 14.37 (20.49) | 10.96 (23.06)

28. Secondary Outcome: Mean Change From Baseline in 36-Item Short Form Health Survey of Quality of Life at Weeks 12, 24, 52, and 104
Description: The 36-Item Short Form Health Survey (SF-36) is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical Component Summary (PCS) and Mental Component Summary (MCS) measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 72 | 73 | 79
Scores on a scale
  PCS Week 12, n=72, 73, 79 | 11.2 (13.4) | 14.2 (14.0) | 6.8 (14.1)
  MCS Week 12, n=72, 71, 7 | 6.2 (12.3) | 10.9 (14.1) | 3.9 (12.7)
  PCS Week 24, n= 72, 74, 76 | 16.3 (15.4) | 13.6 (16.4) | 9.1 (15.1)
  MCS Week 24, n=67, 72,75 | 9.5 (13.6) | 9.3 (16.6) | 5.7 (13.9)
  PCS Week 52, n=62, 63, 68 | 18.9 (16.0) | 20.1 (17.2) | 15.7 (17.0)
  MCS Week 52, n=61, 63, 69 | 10.1 (12.9) | 13.6 (15.8) | 10.3 (16.6)
  PCS Week 104, n=52, 57, 60 | 15.2 (19.8) | 15.1 (18.3) | 13.9 (19.9)
  MCS Week 104, n=51, 57, 60 | 9.4 (12.2) | 9.7 (16.5) | 8.6 (15.5)

29. Secondary Outcome: Mean Change From Baseline in Patient Global Health Visual Analog Scale Score of Quality of Life at Weeks 12, 24, 52, and 104
Description: Patient global health VAS score ranges from 0 to 100 and a higher score indicates worse QoL. Patient global health VAS is a component of DAS28.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 101 | 99 | 103
Scores on a scale
  Week 12, n=101, 99, 103 | -25.8 (25.7) | -24.2 (24.7) | -14.8 (25.4)
  Week 24, n= 97, 95, 96 | -33.9 (23.5) | -29.2 (26.1) | -20.4 (27.3)
  Week 52, n=84, 90, 84 | -34.3 (26.1) | -34.9 (26.2) | -31.5 (28.3)
  Week 104, n=76, 83, 74 | -33.2 (22.1) | -34.3 (27.4) | -36.2 (28.6)

30. Secondary Outcome: Mean Change From Baseline in Physician Global Health Visual Analog Scale Score of Quality of Life at Weeks 12, 24, 52, and 104
Description: Physician global health VAS score ranges from 0 to 100 and a higher score indicates worse QoL. Physician global health VAS is a component of DAS28.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 79 | 82 | 79
Scores on a scale
  Week 12, n=79, 82, 79 | -35.4 (23.0) | -34.6 (23.1) | -23.0 (23.1)
  Week 24, n=74, 75, 78 | -43.9 (25.1) | -43.8 (21.1) | -31.0 (25.7)
  Week 52, n=71, 71, 71 | -45.4 (24.9) | -46.9 (23.3) | -37.7 (23.5)
  Week 104, n=61, 68, 64 | -43.7 (26.6) | -50.7 (23.5) | -41.1 (22.2)

31. Secondary Outcome: Mean Change From Baseline in Patient Pain Visual Analog Scale Score of Quality of Life at Weeks 12, 24, 52, and 104
Description: Participants assessed their pain using a 0 to 10 horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 and is described as "no pain" and the right-hand extreme equals 10 as "unbearable pain" .The final VAS score will be derived by multiplying the original scores by 10.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 95 | 96 | 101
Scores on a scale
  Week 12, n=95, 96, 101 | -28.7 (28.8) | -29.5 (31.0) | -19.7 (25.5)
  Week 24, n=92, 93, 92 | -36.4 (28.3) | -33.5 (27.4) | -28.0 (26.9)
  Week 52, n=78, 83, 82 | -37.9 (26.1) | -36.6 (27.2) | -38.1 (27.1)
  Week 104, n=73, 80, 72 | -34.0 (26.8) | -36.4 (27.0) | -41.0 (24.5)

32. Secondary Outcome: Mean Change From Baseline in Patient General Wellbeing Visual Analog Scale Score of Quality of Life at Weeks 12, 24, 52, and 104
Description: Participants assessed their general wellbeing using a 0 to 10 horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 and is described as " not active at all " and the right-hand extreme equals 10 as " very active " .The final VAS score will be derived by multiplying the original scores by 10.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 30 | 19 | 19
Scores on a scale
  Week 12, n=30, 19, 19 | -27.3 (24.2) | -31.1 (27.0) | -6.6 (27.0)
  Week 24, n=28, 18, 18 | -36.1 (23.7) | -35.6 (34.0) | -16.1 (24.8)
  Week 52, n=23, 17, 15 | -40.9 (22.5) | -45.6 (25.7) | -26.0 (23.1)
  Week 104, n=23, 16, 19 | -31.1 (22.4) | -38.1 (31.7) | -34.7 (27.3)

33. Secondary Outcome: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue Score of Quality of Life at Weeks 12, 24, 52, and 104
Description: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participants response to the questions (with the exception of 2 negatively stated), the greater the participants fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the participant's health status.
Time Frame: From Baseline (Week 0) to Weeks 12, 24, 52 and 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 98 | 98 | 99
Scores on a scale
  Week 12, n=98, 98, 99 | 4.3 (8.9) | 6.5 (8.9) | 3.4 (9.5)
  Week 24, n=98, 99, 94 | 7.3 (9.3) | 6.7 (10.6) | 4.4 (8.5)
  Week 52, n=84, 86, 85 | 6.9 (10.6) | 7.9 (10.4) | 6.4 (10.1)
  Week 104, n=74, 78, 74 | 6.3 (9.7) | 5.8 (10.5) | 7.0 (10.7)

34. Secondary Outcome: Mean Change From Baseline in The Revised Illness Perception Questionnaire (IPQ-R) Score of Quality of Life at Week 12
Description: The IPQ-R includes 9 domains (identity, acute or chronic timeline, consequences, personal and treatment control, illness coherence, timeline cyclical, emotional representations, and cause). For first 8 domains it scores as: 1(strongly disagree), 2(disagree), 3(neither agree/disagree), 4(agree), and 5(strongly agree), except identity as 1(yes) and 0(no). The sum of scores for identity, timeline, consequences, and cyclical domains are ranged from 0-16. High score represent strongly held beliefs about the number of symptoms attributed to RA, the chronicity of the condition, the negative consequences of the illness and the cyclical nature of the condition. The sum of scores for personal and treatment control, coherence dimensions, and emotional representations are ranged from 0-15. High score represent positive beliefs about the number of controllability of RA and a personal understanding of the condition. The data for 'Cause' domain was not considered for analysis in this study.
Time Frame: From Baseline (Week 0) to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 98 | 98 | 99
Scores on a scale
  Identity, n=98, 98, 99 | -0.6 (2.0) | -0.8 (1.8) | -0.1 (2.3)
  Acute or Chronic Timeline, n=95, 97, 92 | -0.1 (0.7) | -0.0 (0.6) | 0.0 (0.5)
  Consequences, n=95, 96, 95 | -0.4 (0.7) | -0.4 (0.7) | -0.2 (0.5)
  Personal Control, n=98, 98, 98 | 0.1 (0.5) | 0.1 (0.6) | -0.1 (0.7)
  Treatment Control, n=98, 96, 94 | 0.2 (0.5) | 0.2 (0.5) | 0.1 (0.5)
  Illness Coherence, n=95, 96, 95 | 0.2 (0.7) | 0.3 (0.7) | 0.2 (0.7)
  Timeline Cyclical, n=95, 98, 96 | -0.2 (0.8) | -0.0 (0.7) | -0.2 (0.6)
  Emotional Representation, n=95, 98, 96 | -0.4 (0.8) | -0.6 (0.9) | -0.5 (0.9)

35. Secondary Outcome: Mean Change From Baseline in The IPQ-R Score of Quality of Life at Week 24
Description: as for outcome 34
Time Frame: From Baseline (Week 0) to Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 98 | 99 | 94
Scores on a scale
  Identity, n=98, 99, 94 | -1.2 (2.1) | -1.0 (1.9) | -0.3 (2.1)
  Acute or Chronic Timeline, n=97, 96, 87 | -0.0 (0.7) | 0.1 (0.6) | 0.0 (0.6)
  Consequences, n=97, 96, 89 | -0.5 (0.7) | -0.4 (0.8) | -0.3 (0.7)
  Personal Control, n=98, 97, 94 | 0.1 (0.6) | 0.0 (0.7) | -0.1 (0.8)
  Treatment Control, n=98, 95, 91, | 0.1 (0.5) | 0.1 (0.5) | 0.2 (0.5)
  Illness Coherence, n=96, 94, 89 | 0.3 (0.7) | 0.3 (0.7) | 0.2 (0.2)
  Timeline Cyclical, n=96, 97,90 | -0.3 (0.7) | -0.2 (0.8) | -0.2 (0.7)
  Emotional Representation, n=96, 97, 90 | -0.5 (0.9) | -0.5 (1.0) | -0.5 (1.0)

36. Secondary Outcome: Mean Change From Baseline in The IPQ-R Score of Quality of Life at Week 52
Description: as for outcome 34
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 84 | 86 | 85
Scores on a scale
  Identity, n=84, 86, 85 | -1.0 (2.3) | -1.4 (2.5) | -1.0 (2.0)
  Acute or Chronic Timeline, n=83, 82, 83 | -0.1 (0.9) | 0.1 (0.7) | 0.1 (0.6)
  Consequences, n=83, 82, 84 | -0.7 (0.9) | -0.7 (0.7) | -0.5 (0.7)
  Personal Control, n=84, 84, 84 | 0.1 (0.6) | 0.1 (0.6) | 0.0 (0.6)
  Treatment Control, n=84, 84, 84 | 0.1 (0.6) | 0.2 (0.6) | 0.2 (0.5)
  Illness Coherence, n=83, 80, 83 | 0.3 (0.7) | 0.4 (0.7) | 0.4 (0.7)
  Timeline Cyclical, n=83, 83, 83 | -0.2 (0.8) | -0.3 (0.8) | -0.3 (0.7)
  Emotional Representation, n=83, 82, 83 | -0.7 (1.0) | -0.7 (1.1) | -0.7 (1.1)

37. Secondary Outcome: Mean Change From Baseline in The IPQ-R Score of Quality of Life at Week 104
Description: as for outcome 34
Time Frame: From Baseline (Week 0) to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 74 | 78 | 74
Scores on a scale
  Identity, n=74, 78, 74 | -1.0 (2.3) | -1.3 (2.1) | -0.9 (2.3)
  Acute or Chronic Timeline, n=69, 75, 72 | 0.0 (0.9) | 0.3 (0.9) | 0.3 (0.7)
  Consequences, n=69, 76, 73 | -0.6 (0.8) | -0.5 (0.8) | -0.5 (0.8)
  Personal Control, n=74, 77, 74 | 0.1 (0.7) | 0.0 (0.7) | 0.0 (0.7)
  Treatment Control, n=72, 76, 73 | 0.1 (0.6) | 0.1 (0.7) | -0.0 (0.7)
  Illness Coherence, n=69, 75,72 | 0.3 (0.7) | 0.4 (0.7) | 0.4 (0.8)
  Timeline Cyclical, n=69, 77, 73 | -0.1 (0.7) | -0.1 (0.8) | -0.1 (0.8)
  Emotional Representation, n=69, 77, 73 | -0.6 (1.0) | -0.7 (1.1) | -0.7 (1.0)

38. Secondary Outcome: Number of Participants With Any Adverse Events, Any Serious Adverse Events, and Adverse Events Leading to Discontinuation
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. A serious adverse event is defined as any event which was fatal (resulted in death), lifethreatening (with immediate risk of death), resulted in a new or prolongation of a current hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, considered medically significant by the investigator, required intervention to prevent one or more of the outcomes listed above.
Time Frame: Up to Week 104
Population: The safety population consisted of all participants who received at least one dose of TCZ/placebo infusion or MTX/placebo capsule and have at least one post-baseline safety assessment.
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 106 | 103 | 108
Number of participants
  Any AE | 105 | 99 | 106
  Any SAE | 16 | 19 | 13
  AEs Leading to Discontinuation | 23 | 16 | 19

39. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values at Week 12
Description: Laboratory parameters included hematology, chemistry and lipids. Any treatment-emergent abnormal laboratory result accompanied by clinical symptoms or leading to a change in study medication or requiring a change in concomitant therapy was considered clinically significant. Participants with clinically significant laboratory values are reported in the below table.
Time Frame: Week 12
Population: The safety population consisted of all participants who received at least one dose of TCZ/placebo infusion or MTX/placebo capsule and have at least one post-baseline safety assessment. n = number of participants evaluable at particular time of assessment.
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 104 | 101 | 100
Number of participants
  Absolute Neutrophil Count, n=97, 94, 97 | 2 | 0 | 0
  Eosinophil, n=93, 90, 93 | 0 | 0 | 0
  Hematocrit, n=104,100,100 | 0 | 0 | 0
  Hemoglobin, n=104, 101,100 | 0 | 0 | 1
  Red blood cells, n=104,100,100 | 1 | 0 | 0
  Thrombocyte, n=104, 101,100 | 0 | 0 | 0
  White blood cells, n=104, 101,100 | 3 | 2 | 0
  Alkaline phosphatase, n=104,101, 99 | 0 | 0 | 0
  Alanine transaminase (ALT), n=104, 101,100 | 4 | 2 | 2
  Aspartate aminotransferase (AST), n=104,100,100 | 1 | 1 | 1
  Creatinine, n=104,101,100 | 1 | 0 | 0
  CRP, n=103,100,100 | 3 | 0 | 2
  High-density lipoprotein (HDL), n=101,100,99 | 1 | 0 | 1
  Low-density lipoprotein (LDL), n=99,97,98 | 5 | 2 | 2
  Total cholesterol, n=102,100,99 | 7 | 5 | 2
  Triglycerides, n=102,100, 99 | 2 | 2 | 2

40. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values at Week 24
Description: as for outcome 39
Time Frame: Week 24
Population: as for outcome 39
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 100 | 101 | 98
Number of participants
  Absolute Neutrophil Count, n=96, 97 ,97 | 1 | 0 | 0
  Eosinophil, n=91, 93, 93 | 0 | 0 | 0
  Hematocrit, n=100, 99, 98 | 0 | 1 | 0
  Hemoglobin, n=100, 100, 98 | 0 | 1 | 1
  RBC, n=99, 100, 98 | 0 | 1 | 0
  Thrombocyte, n=100, 100, 98 | 0 | 0 | 0
  WBC, n=100, 101, 98 | 2 | 0 | 0
  Alkaline phosphatase, n=100, 101, 98 | 0 | 0 | 0
  ALT, n=100, 101, 98 | 2 | 2 | 5
  AST, n=100, 101, 98 | 2 | 0 | 1
  Creatinine, n=100, 101, 98 | 0 | 0 | 0
  CRP, n=100, 101, 97 | 0 | 0 | 2

41. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values at Week 52
Description: as for outcome 39
Time Frame: Week 52
Population: as for outcome 39
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 86 | 92 | 88
Number of participants
  Absolute Neutrophil Count, n=83, 90, 85 | 0 | 0 | 0
  Eosinophil, n=81, 88, 82 | 0 | 0 | 4
  Hematocrit, n=86, 92, 87 | 0 | 0 | 1
  Hemoglobin, n=86, 92, 88 | 0 | 0 | 2
  RBC, n=86, 91, 87 | 0 | 0 | 1
  Thrombocyte, n=85, 92, 88 | 0 | 0 | 1
  WBC, n=86, 92, 88 | 0 | 1 | 0
  Alkaline phosphatase, n=86, 92, 87 | 0 | 0 | 0
  ALT, n=86, 92, 88 | 0 | 0 | 7
  AST, n=86, 91, 88 | 0 | 0 | 2
  Creatinine, n=86, 92, 88 | 0 | 2 | 0
  CRP, n=86, 91, 87 | 1 | 0 | 0

42. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values at Week 104
Description: as for outcome 39
Time Frame: Week 104
Population: as for outcome 39
Measure: Number; unit: Number of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Number analyzed (Participants) | 78 | 80 | 78
Number of participants
  Absolute Neutrophil Count, n=75, 78, 77 | 0 | 0 | 1
  Eosinophil, n=72, 77, 74 | 0 | 0 | 0
  Hematocrit, n=75, 78, 77 | 1 | 0 | 1
  Hemoglobin, n=78, 80, 78 | 1 | 0 | 1
  RBC, n=76, 79, 77 | 1 | 0 | 0
  Thrombocyte, n=78, 79, 78 | 0 | 1 | 1
  WBC, n=78, 80, 78 | 1 | 0 | 1
  Alkaline phosphatase, n=78, 79, 78 | 0 | 0 | 0
  ALT, n=78, 80, 78 | 0 | 0 | 2
  AST, n=78, 80, 78 | 0 | 0 | 2
  Creatinine, n=78, 79, 78 | 1 | 1 | 0
  CRP, n=78, 80, 78 | 1 | 0 | 0
  HDL, n=76, 76, 72 | 1 | 0 | 1
  LDL, n=74, 74, 72 | 0 | 1 | 3
  Total cholesterol, n=76, 76, 72 | 0 | 2 | 3
  Triglycerides, n=76, 76, 72 | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: Up to Week 104
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Population, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post-baseline.
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo Methotrexate | Methotrexate + Placebo Tocilizumab
Serious Adverse Events (participants affected / at risk) | 16/106 | 19/103 | 13/108
Other Adverse Events (participants affected / at risk) | 105/106 | 99/103 | 106/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab + Methotrexate (N=106) | Tocilizumab + Placebo Methotrexate (N=103) | Methotrexate + Placebo Tocilizumab (N=108)
Pneumonia (Infections and infestations) | 0 | 2 | 2
Bursitis infective (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Viral pericarditis (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 1 | 0
Ill-defined disorder (General disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0
Intervertebral disc operation (Surgical and medical procedures) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab + Methotrexate (N=106) | Tocilizumab + Placebo Methotrexate (N=103) | Methotrexate + Placebo Tocilizumab (N=108)
Nasopharyngitis (Infections and infestations) | 38 | 40 | 37
Influenza (Infections and infestations) | 18 | 13 | 10
Cystitis (Infections and infestations) | 6 | 6 | 11
Oral herpes (Infections and infestations) | 7 | 7 | 6
Urinary tract infection (Infections and infestations) | 6 | 3 | 8
Nausea (Gastrointestinal disorders) | 27 | 20 | 48
Diarrhoea (Gastrointestinal disorders) | 19 | 12 | 20
Mouth ulceration (Gastrointestinal disorders) | 15 | 12 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 12 | 13
Abdominal discomfort (Gastrointestinal disorders) | 6 | 5 | 15
Vomiting (Gastrointestinal disorders) | 4 | 6 | 8
Fatigue (General disorders) | 30 | 25 | 34
Influenza like illness (General disorders) | 6 | 8 | 11
Malaise (General disorders) | 4 | 8 | 9
Oedema peripheral (General disorders) | 8 | 6 | 2
Alanine aminotransferase increased (Investigations) | 25 | 16 | 28
Aspartate aminotransferase increased (Investigations) | 9 | 6 | 15
Headache (Nervous system disorders) | 20 | 15 | 22
Dizziness (Nervous system disorders) | 12 | 12 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 10 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 12 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 12
Bursitis (Musculoskeletal and connective tissue disorders) | 7 | 6 | 6
Leukopenia (Blood and lymphatic system disorders) | 13 | 12 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 9 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 12 | 11
Eczema (Skin and subcutaneous tissue disorders) | 8 | 6 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 5 | 7
Hypertension (Vascular disorders) | 11 | 10 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.